CLINICAL TRIAL: NCT04996134
Title: Domperidone Protocol - FDA Expanded Access Program
Brief Title: Domperidone Expanded Access Treatment Program
Status: No longer available | Type: Expanded Access
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00107013; 17-123 (16-817) (Other: Aurora Baycare Medical Center)
Record Dates: First submitted 2021-08-03; First posted 2021-08-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Domperidone Oral Product — 10-30 mg of oral domperidone administered QID.

SUMMARY:
To allow the use of domperidone by patients with gastrointestinal disorders who have failed standard therapy.

DETAILED DESCRIPTION:
To provide oral domperidone to patients ≥12 years of age where, according to the investigator's judgment, a prokinetic effect is needed for the relief of refractory gastroesophageal reflux disease with upper gastrointestinal (GI) symptoms, gastroparesis, and chronic constipation in patients whom the potential benefit may outweigh the risk of cardiovascular adverse reactions including QT prolongation, Torsades de Pointes, and death.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 12 and older
3. Symptoms or manifestations secondary to GERD (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms), gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation that are refractory to standard therapy.
4. Patients must have a comprehensive evaluation to eliminate other causes of their symptoms.
5. Patient has signed informed consent for the administration of domperidone that informs the patient of potential adverse events

Exclusion Criteria:

History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsades de Pointes. Patients with minor forms of ectopy (PACs) are not necessarily excluded.

1. Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QTc (QTc > 450 milliseconds for males, QTc>470 milliseconds for females).
2. Hepatic dysfunction
3. Renal insufficiency
4. Clinically significant electrolyte disorders.
5. Gastrointestinal hemorrhage or obstruction
6. Presence of a prolactinoma (prolactin-releasing pituitary tumor).
7. Pregnant or breast feeding female
8. Known allergy to domperidone

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John Bosco, MD, Principal Investigator — Aurora BayCare Medical Center
Locations (1):
- Aurora BayCare Medical Center, Green Bay, Wisconsin, United States